CLINICAL TRIAL: NCT06464055
Title: A Phase I/II, Multicenter, Open-Label, Dose-Escalation and Extension Study of GQ1010(an Anti-Trop2 ADC) in Subjects With Advanced Solid Tumors
Brief Title: A Study of GQ1010 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeneQuantum Healthcare (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GQ1010-101
Record Dates: First submitted 2024-06-07; First posted 2024-06-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Advanced Malignant Solid Tumors
MeSH Terms: interventions — Clinical Trials, Phase II as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Dose Escalation (Experimental): GQ1010 will be administered intravenously every 21 days or every 14 days. Dose Escalation will be guided by Bayesian Optimal Interval (BOIN) Design.
  Multiple dose grouping
  Interventions: Drug: Dose Escalation
- Dose Expansion1 (Experimental): GQ1010 at the recommended doses for Expansion (RDEs) . Dose expansion will further evaluate the safety and tolerability in advanced malignant solid tumor subjects.
  Interventions: Drug: Dose Expansion1
- Dose Expansion2 (Experimental): GQ1010 at the recommended doses for Expansion (RDEs). Dose expansion will further evaluate the safety and tolerability in advanced malignant solid tumor subjects.
  Interventions: Drug: Dose Expansion2
- Dose Expansion3 (Experimental): GQ1010 at the recommended doses for Expansion (RDEs) . Dose expansion will further evaluate the safety and tolerability in advanced malignant solid tumor subjects.
  Interventions: Drug: Dose Expansion3
- phase II (Experimental): GQ1010 at the recommended phase II dose (RP2D). Dose expansion will evaluate preliminary efficacy in different types of malignant solid tumor in five cohorts.
  Interventions: Drug: phase II

INTERVENTIONS:
Drug: Dose Escalation — Drug: GQ1010
  Arms: Dose Escalation
Drug: Dose Expansion1 — Drug: GQ1010 dose 1
  Arms: Dose Expansion1
Drug: Dose Expansion2 — Drug: GQ1010 dose 2
  Arms: Dose Expansion2
Drug: Dose Expansion3 — Drug: GQ1010 dose 3
  Arms: Dose Expansion3
Drug: phase II — Drug: GQ1010 RP2D
  Arms: phase II

SUMMARY:
This is an open-label, phase I/II study to evaluate the safety, tolerability, pharmacokinetics and immunogenicity of GQ1010 and preliminary anti-tumor efficacy in advanced malignant solid tumor subjects

DETAILED DESCRIPTION:
This is a Phase 1/2, first in human (FIH), open-label, multicenter study of GQ1010, a Trop-2 directed antibody-drug conjugate (ADC), in participants with previously treated, advanced solid tumors. The study comprises 3 parts: a Phase 1a Dose Escalation, a Phase 1b Dose Expansion, and Phase 2 study. The Phase 1a will investigate the safety and tolerability of GQ1010 and identify one or more recommended doses for expansion (RDEs) and the maximum-tolerated dose (MTD) (if exists). Once the RDEs has been established, Phase 1b will open to identify the recommended phase 2 dose (RP2D) of GQ1010. Then the phase 2 study will open to investigate the preliminary efficacy of GQ1010 in 5 cohorts with different tumor types.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥18 years old.
2. Is able to provide written informed consent and is willing and able to comply with the protocol prior to initiation of any study-related tests or procedures.
3. Has a life expectancy of ≥ 3 months.
4. With histologically or cytologically confirmed locally advanced or metastatic solid malignant tumors with epithelial derived malignancy has relapsed or progressed following local standard treatments, or for which no standard treatment is available. Priority for inclusion but not limited to the following types of cancer: gastric adenocarcinoma/gastroesophageal junction cancer, breast cancer (triple negative and hormone receptor-positive, HER2 negative), colorectal cancer, cholangiocarcinoma, pancreatic cancer, endometrial cancer, ovarian cancer, cervical cancer, etc.
5. Agreed to provide archived tumor tissue specimens (unstained 10 surgical specimens [thickness 4-5μm] was suggested or fresh tissue samples of primary or metastatic sites within 3 years.

   Note: Trop-2 expression was not used to confirm participant eligibility; Tissue samples will be used for subsequent analysis of Trop-2 expression levels and other biomarkers.
6. Measurable tumor lesion based on Response Evaluation Criteria in Solids Tumors (RECIST) version 1.1.
7. Subjects had confirmed disease progression during or after the most recent treatment for locally advanced or metastatic disease, or subjects would not benefit from the former treatment assessed by the investigator .
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. If of reproductive/child-bearing potential(male and female) must agree to use reliable contraceptive measures (include hormonal contraceptives, barrier contraception or abstinence) with their partners during and upon completion of the study and for at least 7 months after the last dose of study drug.
10. Has adequate bone marrow reserve and organ function (no transfusion or hematopoietic-stimulating factor therapy within 14 days):

    * Hemoglobin (HGB) ≥ 9 g/dl
    * Absolute neutrophil count (ANC) ≥ 1,500/mm3,
    * Platelet count (PLT) ≥ 100,000/mm3,.
    * Serum creatinine ≤ 1.5 × ULN or creatinine clearance (Ccr) ≥ 50 ml/min (calculated according to the cockcroft-gault formula),
    * Total bilirubin (TBIL) ≤ 1.5 × ULN (gilbert's syndrome, TBIL ≤ 3 × ULN),
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × ULN (with liver metastases ≤ 5.0 × ULN)
    * International normalized ratio of prothrombin (INR) ≤ 1.5 × ULN, or prothrombin time (PT) ≤ 1.5 × ULN,
    * Activated partial thromboplastin time (APTT) ≤1.5 × ULN. Subjects receiving anticoagulant therapy must have INR and/or APTT≤ the upper limit of the therapeutic range intended for use,
    * Left ventricular ejection fraction ≥50% by echocardiography
11. Has an adequate treatment washout period prior to initial treatment.
12. 3a: Has a pathologically documented HER2 negative (IHC 2+ and ISH* - or ISH unknown, or IHC 1+) advanced/unresectable or metastatic gastric adenocarcinoma/gastroesophageal junction carcinoma(GC/GJC) that relapsed or progressed after standard therapy (at least first-line chemotherapy with or without immune checkpoint inhibitor), or no standard therapy available. Those who relapsed/progressed within 6 months of prior adjuvant/neoadjuvant systemic therapy are not required to receive an additional line of therapy in order to be eligible.
13. 3b: Has a pathologically documented advanced/unresectable or metastatic triple negative breast cancer(TNBC) that relapsed or progressed after standard treatment (at least first-line chemotherapy), or no standard treatment available. Subjects with HER2 low expression who have progressed after treatment with anti-HER2-ADC (such as T-DXd) are admitted.
14. 3b: Has a pathologically documented advanced, or unresectable, or metastatic HER2 negative(IHC2+ with ISH*- or ISH unknown, or IHC1+) HR+BC, is documented refractory or resistant to standard therapy (Was previously treated with a minimum of 1 and a maximum of 4 prior lines of chemotherapy in the advanced/metastatic setting), or no standard therapy available :

    * All subjects must have previously received antitumor endocrine therapy, CDK-4/6 inhibitor therapy, and taxanes;
    * Those who relapsed/progressed within 12 months of prior adjuvant/neoadjuvant systemic therapy are not required to receive an additional line of therapy in order to be eligible.;
    * Subjects with HER2 low expression who have progressed after treatment with anti-HER2-ADC (such as T-DXd) are admitted.
15. 3c: Has a pathologically documented advanced, unresectable, or metastatic colorectal cancer is documented refractory or resistant to standard treatment (at least 2 prior lines systemic therapy, including 5-FU-based chemotherapy and anti-VEGF or anti-EGFR-mAb therapy), or no standard therapy available.

    • Has not progressed or relapsed within 3 months of therapy with irinotecan.
16. 3d: Has a pathologically documented advanced/unresectable or metastatic cervical cancer or endometrial cancer that relapsed or progressed after standard therapy (at least first-line chemotherapy with or without immune checkpoint inhibitor), or no standard therapy available.
17. 3d: Pathologically documented unresectable or metastatic platinum-resistant ovarian cancer that has relapsed or progressed within 6 months of platinum-based chemotherapy, or no standard therapy available. .
18. 3d: Pathologically documented unresectable or metastatic platinum-sensitive ovarian cancer that has relapsed or progressed at least 6 months after the most recent platinum-based chemotherapy , or no standard therapy available. .
19. 3e: Has a pathologically documented advanced/unresectable or metastatic Biliary tract carcinoma(BTC) that relapsed or progressed after standard therapy (at least first-line chemotherapy with or without immune checkpoint inhibitor), or no standard therapy available.
20. 3e: Has a pathologically documented unresectable or metastatic Head and neck squamous cell carcinoma(HNSCC) that relapsed or progressed after at least 1 prior lines of therapy including chemotherapy and ICI or EGFR mAb (in combination or sequential ), or no standard therapy available.
21. 3e: Has a pathologically documented unresectable or metastatic pancreatic cancer that relapsed or progressed after least 1 prior line of systemic therapy, or no standard therapy available. Those who relapsed/progressed within 6 months of prior adjuvant/neoadjuvant systemic therapy are not required to receive an additional line of therapy in order to be eligible. And has not progressed or relapsed within 3 months of therapy with irinotecan.

Exclusion Criteria:

1. Is a lactating mother or pregnant as confirmed by pregnancy tests;
2. Clinically significant concurrent diseases, including but not limited to:

   * Heart failure with New York Heart Association [NYHA] Grade II to IV
   * Myocardial infarction, unstable angina pectoris, or stroke within 6 months prior to the first dose of study drug
   * Newly diagnosed thromboembolic events requiring therapeutic intervention within 6 months prior to the first dose of study drug
   * Severe aortic stenosis
   * Uncontrolled arrhythmia
   * Congenital long QT syndrome
   * Prolonged QT interval (QTcF) as corrected by Fredericia > 470 msec according to 12-lead ECG
   * Uncontrolled hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥110 mmHg) or diabetes (HbA1c ≥9.0%)
   * Clinically significant active infection requiring systemic antibiotic, antiviral, or antifungal treatment
   * Poorly controlled pleural effusion, pericardial effusion, or ascites with clinical symptoms requiring drainage (poorly controlled as carrying a drainage tube or drainage frequency ≥1 / week).;
3. Clinically active brain metastases, defined as untreated and symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms. Has leptomeningeal carcinomatosis, has brain stem metastasis, spinal cord compression. A minimum of 4 weeks must have elapsed between the end of whole brain surgery and study enrollment. Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with steroids may be included in the study if they have recovered from the acute toxic effect of chemotherapy or radiotherapy.
4. Subjects have had other primary malignancies within the last 3 years (other than sufficiently resected non-melanoma skin cancer, cured in situ disease, cured other solid tumors, and/or contralateral breast cancer).
5. Has a history of or currently have interstitial lung disease (including but not limited to pulmonary fibrosis, radiation pneumonia) that requires steroids, or cannot be ruled out by imaging; Patients who currently have active pneumonia or pulmonary function tests that confirm severe impairment of lung function, and patients who require oxygen inhalation.
6. Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder (ie, pulmonary emboli within 3 months of the study enrollment, severe asthma, severe COPD, restrictive lung disease, pleural effusion etc.), or any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (ie, Rheumatoid arthritis, Sjögren's, sarcoidosis etc.), or prior pneumonectomy.
7. Participants who are active or have a clear history of inflammatory bowel disease, or who have esophageal and gastric varices, gastrointestinal obstruction, severe ulcers, gastrointestinal perforation, abdominal abscess, or acute gastrointestinal bleeding within 6 months prior to the first dose of study drug;
8. Imaging (CT or MRI) confirmed that the tumor surrounds important blood vessels or the investigator determines that the tumor is highly likely to invade important blood vessels and cause fatal massive bleeding during subsequent studies;
9. Has an active hepatitis C (HCV antibody positive with HCV RNA above the reference limit) or hepatitis B virus infection (e.g., hepatitis B surface antigen [HBsAg] positive with HBV DNA≥2000 IU/mL); tuberculosis (evidence of active TB infection within 1 year), syphilis (positive for both specific and non-specific antibodies to treponema pallidum); people infected with human immunodeficiency virus (HIV positive).
10. Grade 2 or above corneal disease with clinical symptoms.
11. Previously received Trop-2 targeted therapy, including Trop-2 ADC.
12. Previously received ADC therapy with topoisomerase I inhibitors as payload (HR+HER2-BC and TNBC cohort excepted).
13. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia, chemotherapy-induced grade 2 neuropathy, endocrinopathies which can be well controlled by hormone replacement therapy and other toxicities that remained grade 2 but chronically stable evaluated by the investigator ) not yet resolved to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0, Grade ≤1 or baseline.
14. Has a history of severe hypersensitivity reactions to either the drug substances or inactive ingredients of GQ1010. Has a history of severe hypersensitivity reaction to other monoclonal antibodies.
15. Has any other past or current evidence of any concomitant disease, treatment, or laboratory test abnormality that would increase the safety risk to the subject or interfere with participation of the subject or evaluation of the clinical study in the opinion of the investigator.
16. Nucleic acid test positive for acute severe respiratory syndrome coronavirus type 2 (SARS-CoV-2) within 30 days prior to the first administration of the study drug.
17. Administered live vaccine within 30 days prior to the first administration of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2028-05-23 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase I/II: Incidence and Severity of Adverse Events (AEs) | Screening up to study completion, an average of 1 year
  Incidence and severity of Treatment-emergent adverse events, treatment-related adverse events and serious adverse events, according to NCI-CTCAE Version 5.0 (The number of participants who had treatment-related side effects in population who had received one therapy at least).
  Incidence and severity of TEAEs, TRAE and SAE
Phase Ia: Dose Limiting Toxicities (DLTs) | 21 days or 28 days
  Adverse events will be assessed using NCI CTCAE version 5.0 and will be evaluated by the investigator and the sponsor for the eligibility of DLT.
Phase Ia: Maximal Tolerance Dose (MTD) or recommended doses for dose expansion (RDEs) | After each cohort completes the DLT observation period or has a DLT or becomes not DLT-evaluable
  The SRC will determine the MTD/RDEs based on the totality of data for all tested dose levels.
Phase Ib: Recommended phase II dose (RP2D) | After each cohort completes the safety and efficacy evaluation, an average of 6 months
  The SRC will also determine the RP2D based on the totality and efficacy of data for all tested dose levels.
Phase II: Objective response rate (ORR) determined by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Screening up to study completion, an average of 1 year
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). ORR is evaluated by the number of participants with best overall response of CR and PR.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of GQ1010 | Screening up to study completion, an average of 1 year
  The pharmacokinetics(PK) profile of GQ1010
Time of peak plasma concentration (Tmax) | Screening up to study completion, an average of 1 year
  The pharmacokinetics(PK) profile of GQ1010
Area under the plasma concentration time curve (AUC) of GQ1010 | Screening up to study completion, an average of 1 year
  The pharmacokinetics(PK) profile of GQ1010
Terminal half-life (T1/2) of GQ1010 | creening up to study completion, an average of 1 year
  The pharmacokinetics(PK) profile of GQ1010
Objective response rate (ORR) determined by investigators according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Screening up to study completion, an average of 1 year
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). ORR is evaluated by the number of participants with best overall response of CR and PR (Confirmed CR/PR assessment require at least 1 repeat).
Duration of response (DOR) determined by investigators according to RECIST 1.1 | Screening up to study completion, an average of 1 year
  DoR was defined as the period from the first occurrence of CR or PR to PD or death from any cause. If no PD or death after CR/PR, the cut-off date of progression-free survival (PFS) would be used [Confirmed CR/PR assessment require at least one repeat (≥4 weeks)].
Disease control rate (DCR) determined by investigators according to RECIST 1.1 | Screening up to study completion, an average of 1 year
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). DCR was evaluated by the number of participants with best overall response of CR, PR and stable disease (SD).
Progression-free survival (PFS) determined by investigators according to RECIST 1.1 | Screening up to study completion, an average of 1 year
  Objective tumor response for target lesions will be assessed by imaging/measurement compared with the overall tumor burden at baseline (Day -28 to -1). PFS was defined as the time from first dose to PD or death from any cause.
Overall survival (OS) (only in dose expansion stage) | Screening up to study completion, an average of 1 year
  OS was defined as the time from first dose to death from any cause.
Immunogenicity (anti-drug antibody ADA) | Screening up to study completion, an average of 1 year
  Percentage of subjects producing detectable anti-drug antibodies (ADA)

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Department of Gastrointestinal Oncology, Key Laboratory of Carcinogenesis and Translational Research (Ministry of Education/Beijing), Peking University Cancer Hospital & Institute, Beijing
  - Department of Medical Oncology, Harbin Medical University Cancer Hospital, Harbin
  - Tianjin medical university cancer institute & hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou